CLINICAL TRIAL: NCT03529045
Title: CORE-VNS: Comprehensive Outcomes Registry in Subjects With Epilepsy Treated With Vagus Nerve Stimulation Therapy
Brief Title: Registry of Subjects With Drug Resistant Epilepsy and Treated With the VNS Therapy System.
Acronym: CORE-VNS
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: LNN-801
Record Dates: First submitted 2018-02-22; First posted 2018-05-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy; Seizures; Drug Resistant Epilepsy
Keywords: VNS; VNS Therapy; Vagus Nerve Stimulation
MeSH Terms: conditions — Epilepsy; Seizures; Drug Resistant Epilepsy | interventions — Vagus Nerve Stimulation; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- VNS Therapy: Any approved VNS Therapy System (according to local regulations) may be used in this registry.
  Interventions: Device: Vagus Nerve Stimulation (VNS) Therapy

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) Therapy — The VNS Therapy System is a commercially available device that will be used by licensed medical practitioners trained in the use of VNS Therapy, per the practitioners' medical judgement.

SUMMARY:
Multicenter global post-market registry of subjects diagnosed with drug resistant epilepsy and treated with the VNS Therapy System.

DETAILED DESCRIPTION:
The purpose of this registry is to evaluate clinical outcome and safety data in subjects with drug resistant epilepsy treated with the VNS Therapy System. The study will collect outcomes for subjects treated with VNS Therapy in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of drug resistant epilepsy treated with VNS Therapy. Eligible subjects include those not previously treated with VNS Therapy as well as subjects receiving replacement generators.
* Able and willing to comply with the frequency of study visits.
* Subject, or legal guardian, understands study procedures and voluntarily signs an informed consent in accordance with institutional policies. In the event that the subject is under the age of 18, the subject may also be required (per EC/IRB) to sign an assent affirming their agreement to participate.

Exclusion Criteria:

• There are no exclusion criteria in this study. Investigators should refer to the local instructions for use for VNS Therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with drug resistant epilepsy and treated with the VNS Therapy System. Eligible subjects include those receiving VNS Therapy for the first time, as well as those that are being re-implanted with VNS
Sampling Method: Non-Probability Sample
Enrollment: 827 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Seizure Frequency | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  The average seizure frequency per month over the last 3 months (by type) will be collected
Maximum Seizure Free Period | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  The maximum seizure free period over the last 3 months will be collected
Seizure Severity | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  Seizure severity is a categorical outcome and will be rated by the subject using the following categories: Very mild, Mild, Moderate, Severe, Very Severe
Post-ictal Severity | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  Seizure severity is a categorical outcome and will be rated by the subject using the following categories: Very mild, Mild, Moderate, Severe, Very Severe
Change in Quality of Life | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  Quality of life is a categorical outcome and will be rated by the subject using the following categories: Very good: could hardly be better, Pretty good, Good and bad parts about equal, Pretty bad, Very bad: could hardly be worse
Quality of Sleep | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  Quality of sleep will be reported using the Pittsburgh Sleep Quality Index for subjects 18 years and older and using the Children's Sleep Habit Questionnaire for subjects 2-17 years old; quality of sleep will not be assessed in children under 2 years old
Anti-epileptic Drug Use | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  The name and dose of anti-epileptic drugs used will be collected on a case report form
Rescue Drug Use | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  The number of times a rescue drug was used will be collected
Seizure Related Emergency Department Visits | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  The number of times a patient had a seizure related emergency department (ED) visit will be collected
Seizure Related Hospitalizations | Baseline, 3, 6, 12, 24, and 36 months after implant; long term follow-up data through 60 months may be collected, if applicable
  The number of times a patient had a seizure related inpatient hospitalization and the length of each stay will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Way, Study Director — LivaNova, Inc.
Locations (62):
- United States (19):
  - St. Mary's Hospital, Grand Junction, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Research Institute of Orlando, Orlando, Florida
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Via Christi Health, Wichita, Kansas
  - Tulane University, New Orleans, Louisiana
  - Dent Neurosciences Research Center, Amherst, New York
  - State University of New York, Syracuse, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Neurology Associates, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Child Neurology Consultants of Austin, Austin, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Valley Health System, Winchester, Virginia
  - Ascension Columbia St. Mary's Hospital, Milwaukee, Wisconsin
- Australia (5):
  - Queensland Children's hospital, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Royal Children's hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Kepler Universitätsklinikum, Linz, Austria
- Belgium (2):
  - UCL Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Brazil (2):
  - Fundação Felice Rosso, Hospital Felício Rocho, Belo Horizonte
  - Instituto Estadual do Cérebro Paulo Niemeyer, Rio de Janeiro
- Canada (5):
  - London Health Sciences Centre Research Inc., London, Ontario
  - London Health Sciences Centre Research Inc. (London Victoria), London, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
- China (3):
  - Sanbo Brain Hospital Capital Medical University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Guangzhou Women and Children's Medical Center, Guangzhou
- India (3):
  - P.D. Hinduja National Hospital, Mumbai, Maharashra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - St.-John Medical College and Hospital, Bangalore
- Israel (3):
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Ospedale Bellaria, Bologna
  - Bambino Gesu Pediatric Hospital, Rome
- Japan (3):
  - National Center Hospital of Neurology and Psychiatry, Kodaira
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - The University of Tokyo Hospital, Tokyo
- Netherlands (3):
  - Kempenhaeghe, Heeze
  - Sophia Kinderziekenhuis, Rotterdam
  - Stichting Epilepsie Instellingen Nederland (SEIN), Zwolle
- Poland (2):
  - University Clinical Center, Katowice
  - Children's Memorial Health Institute, Warsaw
- Centro Hospitalar de São João, Porto, Portugal
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Jeddah
  - King Faisal Specialist Hospital & Research Center, Riyadh
- United Kingdom (6):
  - Southmead Hospital, Bristol
  - King's College Hospital, London
  - Royal Victoria Infirmary Hospital, Newcastle upon Tyne
  - Norfolk and Norwich Hospitals NHS Foundation Trust, Norwich
  - John Radcliffe Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Ekinci O, Isik U, Gunes S, Ekinci N. Understanding sleep problems in children with epilepsy: Associations with quality of life, Attention-Deficit Hyperactivity Disorder and maternal emotional symptoms. Seizure. 2016 Aug;40:108-13. doi: 10.1016/j.seizure.2016.06.011. Epub 2016 Jun 27. PMID 27394056
- [Background] Goodlin-Jones BL, Sitnick SL, Tang K, Liu J, Anders TF. The Children's Sleep Habits Questionnaire in toddlers and preschool children. J Dev Behav Pediatr. 2008 Apr;29(2):82-88. doi: 10.1097/dbp.0b013e318163c39a. PMID 18478627
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Result] Sen A, Verner R, Valeriano JP, Lee R, Zafar M, Thomas R, Kotulska K, Jespers E, Dibue M, Kwan P; CORE-VNS Registry Group. Vagus nerve stimulation therapy in people with drug-resistant epilepsy (CORE-VNS): rationale and design of a real-world post-market comprehensive outcomes registry. BMJ Neurol Open. 2021 Dec 23;3(2):e000218. doi: 10.1136/bmjno-2021-000218. eCollection 2021. PMID 35018342
- [Result] Kwan P, Boffini M, Fahoum F, El Tahry R, O'Brien TJ, Keough K, Boggs J, Goldberg-Stern H, Beraldi F, Giannicola G, Lee YC, Sen A; CORE-VNS Registry Group. Baseline characteristics and predictors for early implantation of vagus nerve stimulation therapy in people with drug-resistant epilepsy: Observations from an international prospective outcomes registry (CORE-VNS). Epilepsia Open. 2024 Oct;9(5):1837-1846. doi: 10.1002/epi4.13015. Epub 2024 Aug 24. PMID 39180426